CLINICAL TRIAL: NCT00615719
Title: Utility of 64-slice Multidetector CT Coronary Angiography in the Evaluation of Low to Intermediate Risk ED Patients
Brief Title: Computed Tomographic Coronary Angiography for Acute Chest Pain Evaluation
Acronym: EDCCTA
Status: Terminated | Type: Observational
Why Stopped: Enrollment rate was too slow.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 20061756; PT101207 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2007-12-25; First posted 2008-02-14 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Acute Coronary Syndromes; Coronary Artery Disease
Keywords: Chest Pain; Coronary Angiography; Acute Coronary Syndromes; Computed Tomography
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED patients undergoing coronary CTA: Emergency Department patients suspected of having acute coronary syndrome undergoing Coronary Computed Tomographic angiography.

SUMMARY:
The purpose of this study is to evaluate whether 64-slice Computed Tomographic coronary angiography is useful for rapid diagnosis or exclusion of significant coronary artery disease in patients who present to the Emergency Department with chest pain.

DETAILED DESCRIPTION:
The acute coronary syndromes (ACS), which encompass unstable angina (UA) and both ST elevation and non-ST elevation myocardial infarction (STEMI and non-STEMI), are the leading cause of death in the United States. In addition, they account for a significant number of hospital admissions (300,000 per year for STEMI, >1,000,000 per year for non-ST elevation ACS). Differentiation of patients with ACS from those with chest pain due to other causes, as well as risk stratification of those within the ACS group, are critically important.

In the Emergency Department(ED), the ECG is initially used to distinguish patients with STEMI from those with non-STEMI and other ACS. Subsequent workup in non-STEMI patients is aimed at rapidly distinguishing those who require admission and possible intervention or intensive medical therapy, from those who can be safely discharged. However, because of the frequent inability to determine whether symptoms are related to an ACS during this initial ED visit, further evaluation is often needed, resulting in an estimated 5,000,000 admissions per year.

Currently, a variety of modalities are used in this process of risk stratification, with resting myocardial perfusion imaging (MPI) often assuming a central role. This modality has an overall sensitivity of 80% and an excellent negative predictive value (95-97%). Resting MPI therefore enables clinicians to safely triage low risk patients to delayed stress testing or discharge. However, as with any test, this technique has limitations, including an increased incidence of equivocal findings in obese patients, lower sensitivity in patients without ongoing symptoms, and unsuitability in patients with previous myocardial damage. Perhaps most importantly, alternative diagnoses such as aortic dissection or pulmonary embolism cannot be evaluated with myocardial perfusion imaging.

If coronary Computed Tomographic angiography (CTA) could be shown to be a robust technique in the clinical setting, it could become a powerful tool in the triage of patients with ACS. Computed Tomography (CT) of the chest is currently considered the gold standard for evaluation of the two most common serious alternative chest pain diagnoses - aortic dissection and pulmonary embolism. A single, rapid comprehensive imaging study that could reliably diagnose or exclude coronary artery disease, aortic dissection, and pulmonary embolism would allow quicker and more appropriate triage of this acutely ill population.

However, in keeping with the principles of evidence-based medicine, before comprehensive gated chest CT angiography can be recommended in preference to existing techniques, systematic comparative studies should be performed. In this study, the results of the CTA will be compared with those of the resting MPI, which is part of the standard ED evaluation of chest pain at this institution. In addition, a majority of these patients subsequently undergo stress MPI. It is therefore anticipated that the stress MPI results will also be compared with the CTA findings.

ELIGIBILITY:
Inclusion Criteria:

* ECG negative for acute MI
* Must be low to intermediate risk for ACS based on the initial ECG, history, and physical, in the absence of ischemic ECG changes and positive markers.
* Must be likely to have stress MPI or coronary arteriography as part of the diagnostic evaluation.

Exclusion Criteria:

* Creatinine > 1.5 mg/dL
* Allergy to radiographic contrast
* Pregnancy
* Contraindication to beta-blocker administration
* Inability to hold breath for 12 seconds
* Inability to place an 18-gauge IV angiocatheter in an antecubital vein
* Arrhythmia that will preclude gating of the CTA
* Prior bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department patients with chest pain considered suspicious for acute coronary syndrome, who were to undergo standard nuclear perfusion imaging as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Grizzard, MD, Principal Investigator — Virginia Commonwealth University; Michael C. Kontos, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU Medical Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ED Patients Undergoing Coronary CTA: Usefulness of Computed Tomographic (CT) Coronary Angiography (CTCA) to Evaluate Emergency Department (ED) Patients With Chest Pain (EDCCTA). Patients were to undergo Coronary CT angiography in addition to the nuclear perfusion imaging performed as the standard of care.
Period: Overall Study
Arm/Group | ED Patients Undergoing Coronary CTA
Started | 35
Completed | 30
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | ED Patients Undergoing Coronary CTA
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: The Presence of Acute Coronary Syndromes(ACS).
Description: The presence of ACS was determined by either cardiac angiography, nuclear perfusion imaging or a clinical course deemed consistent with ACS by final chart review. The number of participants with ACS was determined.
Time Frame: During the presenting illness, usually within two to three days.
Population: Only 30 evaluable patients in study powered for 80 patients.
Measure: Number; unit: participants
Groups:
- Computed Tomographic Coronary Angiography for Chest Pain Evalu: Usefulness of Computed Tomographic (CT) Coronary Angiography (CTCA) to Evaluate Emergency Department (ED) Patients With Chest Pain (EDCCTA)
Arm/Group | Computed Tomographic Coronary Angiography for Chest Pain Evalu
Number analyzed (Participants) | 30
participants | 1

ADVERSE EVENTS:
Arm/Group | ED Patients Undergoing Coronary CTA
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No